CLINICAL TRIAL: NCT02442648
Title: B-Cell Targeted Desensitization With Carfilzomib for Preformed Anti-HLA Antibodies in Patients Awaiting Kidney Transplantation
Brief Title: B-Cell Targeted Carfilzomib Desensitization
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: E. Steve Woodle (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, E. Steve Woodle, Director, Solid Organ Transplantation, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Carfilzomib
Record Dates: First submitted 2015-03-04; First posted 2015-05-13 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Transplants and Implants
Keywords: Renal Transplantation; Carfilzomib; Kyprolis; Desensitization
MeSH Terms: interventions — carfilzomib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A (5-8 patients) - Carfilzomib (Experimental): Two cycles of carfilzomib desensitization given.
  Interventions: Drug: Carfilzomib
- Group B (5-8 patients) - Carfilzomib/plasmapheresis (Experimental): Two cycles of carfilzomib desensitization given with weekly plasmapheresis prior to carfilzomib therapy
  Interventions: Drug: Carfilzomib
- Group C (5-8 patients) - Rituximab/Carfilzomib/plasmapheresis (Experimental): 1 dose of rituximab prior to two cycles of carfilzomib desensitization given with weekly plasmapheresis prior to carfilzomib therapy
  Interventions: Drug: Carfilzomib; Drug: Rituximab
- Group D (5-8 patients) - Rituximab/Carfilzomib/plasmapheresis (Experimental): 1 dose of rituximab prior to three cycles of carfilzomib desensitization given with weekly plasmapheresis prior to carfilzomib therapy
  Interventions: Drug: Carfilzomib; Drug: Rituximab

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib will be administered for desensitization per study protocol.
  Other Names: Krypolis
Drug: Rituximab — Rituximab will be administered for desensitization per study protocol.
  Other Names: Rituxan
  Arms: Group C (5-8 patients) - Rituximab/Carfilzomib/plasmapheresis; Group D (5-8 patients) - Rituximab/Carfilzomib/plasmapheresis

SUMMARY:
The primary purpose of this study is to provide a preliminary evaluation of the safety and potential efficacy of carfilzomib in reducing HLA antibody levels in highly sensitized kidney transplant candidates.

DETAILED DESCRIPTION:
This study is a non-randomized, open label, iterative pilot study. The duration of study will include a 16 month enrollment period and 5 to 6 months of follow-up. A total of 32 patients, male and female, between the ages 18 to 65 will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between 18 and 65 years of age, inclusive.
2. Voluntary written informed consent.
3. Female subject is either postmenopausal for at least 1 year prior to initiation of study treatment, is surgically sterilized, or if of childbearing potential, agrees to practice 2 effective methods of contraception through 3 months after the last dose of carfilzomib.
4. Male subjects, even if surgically sterilized (i.e. status post-vasectomy) must agree to 1 effective contraception.
5. Patient with eligible living donor will have: 1) positive cytotoxic crossmatch, or 2) moderate to strongly positive T or B cell flow cytometry crossmatch (with confirmed donor-specific antibodies (DSAs) on solid-phase assay at screening, or 3) > 2 low to moderate level DSAs (DSA value from 1500 - 8000 MFI).
6. LVEF ≥ 45% within 3 months of evaluation.
7. Patient that is on the kidney transplant waiting list awaiting a deceased donor transplant and has a current or peak cytotoxic or calculated panel reactive antibody (PRA) > 30%.
8. Patient must have no known contraindications to treatment with carfilzomib or rituximab.
9. Review of pre-transplant medical clearance by the patient's dialysis nephrologist or transplant nephrologist or treating physician to assure the patient is medically acceptable for study entry.
10. Patient must be vaccinated against hepatitis B virus.

Exclusion Criteria:

1. Patient has significant neuropathy (Grades 3 - 4, or Grade 2 with pain) by CTCAE criteria within 14 days before enrollment.
2. Myocardial infarction within 6 months prior to enrollment or has ADQI Heart Failure in ESRD Classification System Class 2NR or greater (Appendix B), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
3. Patient has received other investigational drugs within 14 days prior to initiation of study treatment.
4. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
5. Diagnosed or treated for another malignancy within 2 years of enrollment, with the exception of: 1) complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, 2) an in situ malignancy, 3) low-risk prostate cancer after curative therapy, or 4) any cancer with a cure rate ≥ 99%.
6. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies.
7. Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize carfilzomib)
8. Patients with a hemoglobin count <8 g/dL (80 g/L) (subjects may be receiving red blood cell [RBC] transfusions in accordance with institutional guidelines), absolute neutrophil count < 1,000/mm3 or platelet count < 75,000/mm3 within 14 days of consent.
9. Patients who are anti-HIV-positive, or HBsAg-positive, or anti-HCV positive with a detectable HCV viral load on testing performed within one year of consent.
10. Patients with current or recent severe systemic infections requiring treatment (systemic antibiotics, antivirals, or antifungals) within the 2 weeks prior to initiation of study treatment.
11. Receipt of a live vaccine within 4 weeks prior to initiation of study treatment.
12. Evidence of severe liver disease by medical history or physical exam with abnormal liver profile (aspartate aminotransferase [AST], alanine aminotransferase [ALT] or total bilirubin > 1.5 times upper limit of normal [ULN]) on testing performed within 30 days of consent.
13. Female subject is pregnant or breast-feeding.
14. Any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.
15. Patient is not yet on dialysis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2014-12; Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Safety of carfilzomib will be assessed by incidence of grade 3 and above non-hematologic toxicities, incidence of grade 4 hematologic toxicities and incidence of all grades of peripheral neuropathy | 6 months
  The primary objective of the proposed study is to evaluate the safety of carfilzomib alone and in combination with plasmapheresis, with or without rituximab, for desensitization in highly sensitized kidney transplant candidates. Safety will be assessed by overall safety of carfilzomib when used in the desensitization setting, incidence of grade 3 and above non-hematologic toxicities, incidence of grade 4 hematologic toxicities and incidence of all grades of peripheral neuropathy.

SECONDARY OUTCOMES:
Efficacy of carfilzomib | 6 months
  The primary objective of the proposed study is to evaluate the efficacy of carfilzomib alone and in combination with plasmapheresis, with or without rituximab, for desensitization in highly sensitized kidney transplant candidates. Efficacy will be measured by percent reduction in immunodominant DSA (iDSA) [highest titer DSA (MFI)] and/or immunodominant antibody (iAb) from pre-treatment to 48 hours after the last plasmapheresis treatment.

CONTACTS AND LOCATIONS:
Overall Officials: E. Steve Woodle, MD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio